CLINICAL TRIAL: NCT00840138
Title: Comparison of Iatrogenic Common Bile Duct Injuries Following Open Cholecystectomy vs Laparoscopic Cholecystectomy
Brief Title: A Comparison of Bile Duct Injuries Following Open Cholecystectomy Versus Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Ireneusz Kozicki, Medical Centre of Postgraduate Education, Poland
Other Study IDs: Kozicki321
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Cholecystectomy; Common Bile Duct Diseases; Major Bile Duct Injury
MeSH Terms: conditions — Common Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with common bile duct injury after open cholecystectomy
  Interventions: Procedure: Surgical reconstruction
- 2: Patients with common bile duct injury after laparoscopic cholecystectomy
  Interventions: Procedure: Surgical reconstruction

INTERVENTIONS:
Procedure: Surgical reconstruction — Hepaticojejunostomy
  End-to-end anastomosis
  Duct suture over T-tube

SUMMARY:
In this prospective study the investigators compared common bile duct injuries (CBDI) following laparoscopic cholecystectomy (LC) and open cholecystectomy (OC) procedures, 35 patients in each group. To date, no detailed study concerning this matter has been published. LC - CBDI in comparison with OC - CBDI more often concerned young females with a narrow CBD, they were located closer to the liver hilus, and they were more extended.

ELIGIBILITY:
Inclusion Criteria:

* Major common bile duct injury

Exclusion Criteria:

* Minor common bile duct injury

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for common bile duct injuries following laparoscopic and open cholecystectomy procedures.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 1996-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)